CLINICAL TRIAL: NCT06381583
Title: A Liquid Biopsy to Screen for Barrett's Esophagus, Dysplasia, and Esophageal Adenocarcinoma: the EMERALD Multi-center Study.
Brief Title: A Liquid Biopsy for High-risk Pre-cancer Screening of Esophageal Adenocarcinoma
Acronym: EMERALD
Status: Completed | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 23228/EMERALD
Record Dates: First submitted 2024-04-19; First posted 2024-04-24 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Esophagus Cancer; Esophageal Cancer Stage; Esophageal Cancer; Esophageal Neoplasms; Esophagus Adenocarcinoma; Esophagus, Barrett; Barrett Esophagus; Barrett Adenocarcinoma; Barrett Epithelium; Barretts Esophagus With Dysplasia; Barrett's Esophagus Without Dysplasia; Barretts Esophagus With High Grade Dysplasia; Barretts Esophagus With Low Grade Dysplasia; Barrett Esophagus, Long-Segment; Barrett's Esophagus With Dysplasia, Unspecified; Barrett's Esophagus With Esophagitis; Gastroesophageal Reflux; Reflux Disease; Esophageal Adenocarcinoma; Esophageal Dysplasia; Esophageal Neoplasms Malignant
Keywords: Early detection; Micro RNA; miRNA; Liquid biopsy; Dysplasia; Artificial Intelligence; Cancer detection; Long segment Barrett Esophagus; Screening; Surveillance
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (10):
- Patients with Esophageal Adenocarcinoma [Malignant Tissue]: Individuals who underwent endoscopy and were found to only have one of the following:
  * Esophageal adenocarcinoma of any stage
  * Esophageal adenocarcinoma confined to the mucosa (stage Tis)
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Patients with Esophageal Adenocarcinoma [Matching Normal Tissue]: Individuals who underwent endoscopy and were found to only have one of the following:
  * Esophageal adenocarcinoma of any stage
  * Esophageal adenocarcinoma confined to the mucosa (stage Tis)
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Patients with Esophageal Adenocarcinoma or High-Grade Dysplasia Barrett's Esophagus [Test Cohort]: Individuals who underwent endoscopy and were found to only have one of the following:
  * Barrett's Esophagus, with high-grade dysplasia, independently of Barrett's segment length
  * Esophageal adenocarcinoma of any stage
  * Esophageal adenocarcinoma confined to the mucosa (stage Tis)
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Patients with Low-Grade Dysplasia or Long Segment Barrett's Esophagus [Test Cohort]: Individuals who underwent endoscopy and were found to only have Barrett's Esophagus, with one of the following:
  * Craniocaudal maximal extension of 3 cm or more
  * Low-grade dysplasia at most, independently of Barrett's segment length
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Individuals Without Esophageal Adenocarcinoma or Barrett's Esophagus [Test Cohort]: Individuals who underwent endoscopy and were found not to have any Barrett's Esophagus or adenocarcinoma.
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Patients with Esophageal Adenocarcinoma or High-Grade Dysplasia Barrett's Esophagus [Training]: Individuals who underwent endoscopy and were found to only have one of the following:
  * Barrett's Esophagus, with high-grade dysplasia, independently of Barrett's segment length
  * Esophageal adenocarcinoma of any stage
  * Esophageal adenocarcinoma confined to the mucosa (stage Tis)
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Individuals Without Esophageal Adenocarcinoma or Barrett's Esophagus [Training Cohort]: Individuals who underwent endoscopy and were found not to have any Barrett's Esophagus or adenocarcinoma.
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Patients with Esophageal Adenocarcinoma or High-Grade Dysplasia Barrett's Esophagus [Validation]: Individuals who underwent endoscopy and were found to only have one of the following:
  * Barrett's Esophagus, with high-grade dysplasia, independently of Barrett's segment length
  * Esophageal adenocarcinoma of any stage
  * Esophageal adenocarcinoma confined to the mucosa (stage Tis)
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Patients with Low-Grade Dysplasia or Long Segment Barrett's Esophagus [ValidationCohort]: Individuals who underwent endoscopy and were found to only have Barrett's Esophagus, with one of the following:
  * Craniocaudal maximal extension of 3 cm or more
  * Low-grade dysplasia at most, independently of Barrett's segment length
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)
- Individuals Without Esophageal Adenocarcinoma or Barrett's Esophagus [Validation Cohort]: Individuals who underwent endoscopy and were found not to have any Barrett's Esophagus or adenocarcinoma.
  Interventions: Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia)

INTERVENTIONS:
Diagnostic Test: EMERALD (Esophageal MicroRNAs for BaRRett's esophagus, Adenocarcinoma, and Dysplasia) — A panel of circulating microRNA, whose expression level is tested in cell-free derived samples.

SUMMARY:
This study aims to develop a highly sensitive, specific, and cost-effective blood assay for the early detection of esophageal adenocarcinoma and its precursor lesions, using advanced machine learning and state-of-the-art biological analyses.

DETAILED DESCRIPTION:
Esophageal adenocarcinoma (EAC) is a significant global health concern, ranking second in lethality (after pancreatic cancer). Despite being potentially preventable, it remains a leading cause of cancer-related deaths. Traditional screening methods have relied on an endoscopy-first approach to screen for the precursor of EAC, which is Barrett's esophagus (BE). After BE detection, BE is then regularly surveiled to monitor the development of dysplasia, which can be treated to prevent malignant transformation. An endoscopy-first approach is sensitive BE and, therefore, it lowers the risk of developing EAC but it also faces challenges such as invasiveness, cost, and patient compliance.

Non-invasive tests are more appealing to patients than invasive tests and can increase participation rates. Biomarker studies have shown promise, but existing tests lack sensitivity for early-stage EAC and, most importantly, to its precursor lesion BE. This is likely because they over-sampled analytes that are primarily expressed at the EAC end of the spectrum, but not in BE yet during the BE to EAC sequence.

This study proposes developing an innovative liquid biopsy test tailored for EAC and BE to address this. An ideal screening test should be minimally invasive, highly sensitive, and cost-effective. This test would optimize patient compliance and resource allocation by detecting both conditions from a single blood draw. More specifically, circulating microRNA (miRNA) analysis shows promise: tests based on cell-free microRNA (cf-miRNA) have demonstrated high sensitivity.

This study will develop a non-invasive blood test for BE and EAC in four phases:

1. In silico genome-wide profiling of tissue miRNA to select the best candidates for biomarker panels.
2. Prioritization of the biomarkers that are differentially expressed across the entire continuum of BE to EAC sequence, compared to the normal mucosa
3. Transition of these biomarkers to a liquid biopsy assay, confirming their detectability in blood as well as their differential expression in cases compared to controls
4. Utilizing machine learning to identify the most promising candidates and train algorithms for detecting EAC and BE, based on results from quantitative polymerase chain reaction (qPCR) analysis.
5. Independently validating these signatures using diverse cohorts to ensure broad applicability and compare the effectiveness of the blood assay to standard care through retrospective and prospective studies.

This study aims to develop a highly sensitive, specific, and cost-effective liquid biopsy for early detection of BE and EAC. Success could transform clinical practice by preventing EAC through early detection of pre-malignant lesions. Innovations include incorporating pre-malignant lesions into screening. This approach could potentially reduce EAC mortality and incidence and pave the way for new clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* All individuals included in the study need to have had an endoscopic evaluation at the time of blood sampling.
* Received standard diagnostic and staging (as necessary) procedures as per local guidelines, and at least one sample was drawn before receiving any curative-intent treatment.
* Received standard pathological and endoscopic diagnosis and assessment for cohort assignment.

Exclusion Criteria:

* Lack of written informed consent.
* Short segment Barrett's esophagus with no evidence of dysplasia
* Ultra-short segment Barrett's esophagus with no evidence of dysplasia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Four independent cohorts of individuals who belong to one of the following five
  Negative endoscopic findings Barrett's esophagus, at least 3 cm long without low-grade dysplasia (at most) Barrett's esophagus, of any length, with low-grade dysplasia (at most) Barrett's esophagus, of any length, with high-grade dysplasia (at most) Esophageal adenocarcinoma (of any stage, including in situ [Tis]) Colorectal cancer
Sampling Method: Non-Probability Sample
Enrollment: 658 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-04-24 (Actual); Study Completion 2024-04-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Through study completion, an average of 1 year
  True positive rate: the probability of a positive test result, conditioned on the individual truly being positive

SECONDARY OUTCOMES:
Specificity | Through study completion, an average of 1 year
  True negative rate: the probability of a negative test result, conditioned on the individual truly being negative
Proportion of correct predictions (true positives and true negatives) among the total number of cases (i.e., accuracy) | Through study completion, an average of 1 year
  A measure of trueness: proportion of correct predictions (both true positives and true negatives) among the total number of cases examined

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Goel, PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data collected for the study will be made available to others, including de-identified participant data, at publication, via a signed data access agreement and at the discretion of the investigators' approval of the proposed use of such data.

REFERENCES:
- [Derived] Miyoshi J, Mannucci A, Scarpa M, Gao F, Toden S, Whitsett T, Inge LJ, Bremner RM, Takayama T, Cheng Y, Bottiglieri T, Nagtegaal ID, Shrubsole MJ, Zaidi AH, Wang X, Coleman HG, Anderson LA, Meltzer SJ, Goel A; FINBAR-EMERALD collaborative group. Liquid biopsy to identify Barrett's oesophagus, dysplasia and oesophageal adenocarcinoma: the EMERALD multicentre study. Gut. 2025 Jan 17;74(2):169-181. doi: 10.1136/gutjnl-2024-333364. PMID 39562048